CLINICAL TRIAL: NCT04567667
Title: Pharmacokinetics and Metabolism of [14C] BMS-986278 in Healthy Male Participants
Brief Title: Study to Assess the Way the Body Absorbs, Distributes, Breaks Down and Eliminates Radioactive BMS-986278 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IM027-048
Record Dates: First submitted 2020-09-24; First posted 2020-09-28 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-06

CONDITIONS: Healthy Volunteers
Keywords: Healthy volunteers
MeSH Terms: interventions — Sincalide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental)
  Interventions: Drug: [14C] BMS-986278
- Group 2 (Experimental)
  Interventions: Drug: [14C] BMS-986278; Drug: Kinevac®

INTERVENTIONS:
Drug: [14C] BMS-986278 — Specified dose on specified days
Drug: Kinevac® — Specified dose on specified days
  Other Names: Sincalide
  Arms: Group 2

SUMMARY:
The purpose of this study is to assess the way the body absorbs, distributes, breaks down and eliminates radioactive BMS-986278 as well as the safety and tolerability of BMS-986278 in healthy male participants.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* No clinically significant deviation from normal in medical history, physical examination, electrocardiograms (ECGs), vital signs, and clinical laboratory determinations
* Body mass index (BMI) of 18.0 to 30.0 kg/m2, inclusive, and total body weight ≥50 kg (110 lb), at screening. BMI = weight (kg)/(height [m])2
* Males must agree to follow specific methods of contraception, if applicable

Exclusion Criteria:

* Any significant acute or chronic medical condition that presents a potential risk to the participant and/or that may compromise the objectives of the study, including active, or history of, liver disease, or intestinal disorder including irritable bowel syndrome
* Current or recent (within 3 months of study treatment administration) gastrointestinal disease that could impact upon the absorption of study treatment
* Any major surgery within 6 weeks of study treatment administration

Other protocol-defined inclusion/exclusion criteria apply

Ages: 21 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-04-11 (Actual); Study Completion 2021-04-11 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of BMS-986278 | Up to 15 days
Maximum observed plasma concentration (Cmax) of total radioactivity (TRA) | Up to 15 days
Time of maximum observed plasma concentration (Tmax) of BMS-986278 | Up to 15 days
Time of maximum observed plasma concentration (Tmax) of TRA | Up to 15 days
Area under the plasma concentration-time curve extrapolated to infinity (AUC(INF)) of BMS-986278 | Up to 15 days
Area under the plasma concentration-time curve extrapolated to infinity (AUC(INF)) of TRA | Up to 15 days

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to 15 days
Incidence of Serious Adverse Events (AEs) | Up to 73 days
Incidence of clinically significant changes in clinical laboratory results: Hematology tests | Up to 43 days
Incidence of clinically significant changes in clinical laboratory results: Clinical Chemistry tests | Up to 43 days
Incidence of clinically significant changes in clinical laboratory results: Urinalysis tests | Up to 43 days
Incidence of clinically significant changes in vital signs: Blood pressure | Up to 43 days
Incidence of clinically significant changes in vital signs: Heart rate | Up to 43 days
Incidence of clinically significant changes in vital signs: Respiratory rate | Up to 43 days
Incidence of clinically significant changes in vital signs: Body temperature | Up to 43 days
Incidence of clinically significant changes in electrocardiogram (ECG) parameters: QTcF | Up to 43 days
  QTcF = Corrected QT interval using the Fridericia formula. QT interval is the time from the start of the Q wave to the end of the T wave.
Incidence of clinically significant changes in electrocardiogram (ECG) parameters: QT interval | Up to 43 days
  The QT interval is the time from the start of the Q wave to the end of the T wave.
Incidence of clinically significant changes in physical examination findings | Up to 43 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Covance - Clinical Pharmacology Services - Madison, Madison, Wisconsin, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm